CLINICAL TRIAL: NCT04984018
Title: An Single-arm Open-label Phase II Study of Chidamide Plus Camrelizumab as Second-line Therapy for Advanced Esophageal Squamous Cell Carcinoma Treated With PD-1 Blockade.
Brief Title: Chidamide Plus Camrelizumab as Second-line Therapy for Advanced ESCC Treated With PD-1 Blockade
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief Physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WF-001
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide plus Camrelizumab (Experimental): Pts received 200 mg camrelizumab intravenously every 2 weeks and Chidamide 30mg orally twice (biw) per week for 4 consecutive weeks every 6 weeks until disease progression, unacceptable adverse events (AEs) or withdrawal of consent.
  Interventions: Drug: chidamide + camrelizumab

INTERVENTIONS:
Drug: chidamide + camrelizumab — Pts received 200 mg camrelizumab intravenously every 2 weeks and Chidamide 30mg orally twice (biw) per week for 4 consecutive weeks every 6 weeks until disease progression, unacceptable adverse events (AEs) or withdrawal of consent.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of chidamide plus camrelizumab as second-line therapy for advanced esophageal squamous cell carcinoma treated with PD-1 blockade

DETAILED DESCRIPTION:
Although immune checkpoint inhibitors (ICIs) have been tested in esophageal squamous cell carcinoma(ESCC) with demonstrated clinical efficacy，a significant number of patients who have an initial response will develop a secondary resistance and relapse. recent studies on the role of epigenetics in immune evasion have exposed a key role for epigenetic modulators in augmenting the tumour microenvironment and restoring immune recognition and immunogenicity. These discoveries have established a highly promising basis for studies using combined epigenetic and immunotherapeutic agents as anti-cancer therapies. Chidamide is a novel orally active benzamide-type histone deacetylase inhibitor that has shown in vitro activities against a wide array of neoplasms. Hence, the study of chidamide plus camrelizumab as second-line therapy for advanced ESCC treated with PD-1 blockade was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.
2. Age ≥ 18 years on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place).
3. Histologically confirmed diagnosis of ESCC.
4. Have PD after first-line of PD-1 blockade treatment for unresectable, locally advanced, recurrent or metastatic ESCC.
5. Measurable disease per RECIST v1.1 assessed by the local investigator
6. ECOG PS 0 or 1
7. Newly obtained (preferred) or archival tissue sample available
8. Negative urine or serum pregnancy test within 72 h before treatment(females)
9. Willing to use an adequate method of contraception throughout the study and for 120 days after the last dose of study medication and up to 180 days after the last dose of cisplatin
10. Adequate haematologic function, defined as ANC ≥ 1500/μl, platelet count ≥ 100,000/μl and haemoglobin ≥ 9.0 g/dl or ≥5.6 mmol/l
11. Adequate renal function, defined as creatinine ≤ 1.5 × ULN or measured or calculated creatinine clearance ≥ 60 mL/min for those with creatinine levels 1.5 × ULN
12. Adequate hepatic function, defined as total bilirubin ≤1.5 × ULN or direct bilirubin ≤ ULN for those with total bilirubin levels 1.5 × ULN, and ALT/AST levels ≤ 2.5 × ULN
13. Adequate coagulation function, defined as INR ≤ 1.5 × ULN unless the patient is receiving anticoagulant therapy, in which case PT or aPTT should be within the therapeutic range
14. Written informed consent

Exclusion Criteria:

1. Patients with evidence of fistula (either esophageal/bronchial or esophageal/aorta).
2. Evidence of complete esophageal obstruction not amenable to treatment.
3. Active leptomeningeal disease or uncontrolled, untreated brain metastasis.
4. Active autoimmune diseases or history of autoimmune diseases that may relapse
5. Any active malignancy ≤ 2 years before randomization except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
6. Uncontrolled diabetes or > Grade 1 laboratory test abnormalities in potassium, sodium, or corrected calcium despite standard medical management or ≥ Grade 3 hypoalbuminemia ≤ 14 days before treatment.
7. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence within 2 weeks after intervention).
8. History of interstitial lung disease, noninfectious pneumonitis or uncontrolled lung diseases including pulmonary fibrosis, acute lung diseases, etc.
9. Infection (including tuberculosis infection, etc) that requires systemic antibacterial, antifungal or antiviral therapy within 14 days before treatment.
10. A history of severe hypersensitivity reactions to chidamide and monoclonal antibodies.
11. Patients with toxicities (as a result of prior anticancer therapy) that have not recovered to ≤Grade 2 or stabilized, except for AEs not considered a likely safety risk (eg, alopecia, neuropathy, and specific laboratory abnormalities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | up to 2 years
  From date of treatment until the date of death from any cause

SECONDARY OUTCOMES:
ORR | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response(CR+PR)
PFS | up to 1 year
  From date of treatment until the date of first documented progression or date of death from any cause
DOR | up to 1 year
  Refers to the time when the tumor is first evaluated as CR or PR until the first assessment is PD (Progressive Disease) or any cause of death.
DCR | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response and stable response(CR+PR+SD)

OTHER OUTCOMES:
Tumor mutation burden (TMB) | up to 1 year
  Total number of non-synonymous mutations in each coding region of the tumor genome
PD-L1 CPS | up to 1 year
  Number of PD-L1 staining cells (tumor cells)/Total tumor cellsk*100%

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Doctor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University